CLINICAL TRIAL: NCT02439216
Title: A Phase 1/2 Study of Edasalonexent (CAT-1004) in Pediatric Patients With Duchenne Muscular Dystrophy
Brief Title: Phase 1/2 Study in Boys With Duchenne Muscular Dystrophy
Acronym: MoveDMD®
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CAT-1004-201
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Results first posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Muscular Dystrophies; Musculoskeletal Diseases; Nervous System Diseases; Neuromuscular Diseases; Duchenne muscular dystrophy; DMD; dystrophin; dystrophy; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Musculoskeletal Diseases; Nervous System Diseases; Neuromuscular Diseases | interventions — edasalonexent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose 1 (Experimental): Edasalonexent 67 mg/kg/day. Capsules taken by mouth two times per day
  Interventions: Drug: Edasalonexent
- Dose 2 (Experimental): Edasalonexent 100 mg/kg/day. Capsules taken by mouth three times per day
  Interventions: Drug: Edasalonexent
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Edasalonexent
  Other Names: CAT-1004; Edasa
  Arms: Dose 1; Dose 2
Drug: Placebo
  Arms: Placebo

SUMMARY:
The MoveDMD study is a 3-part, Phase 1/2, multi-site study to evaluate the safety, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of edasalonexent (also known as CAT-1004) in pediatric patients with a genetically confirmed diagnosis of DMD. Male patients from ≥4 to <8 years of age will be enrolled.

Edasalonexent is an orally administered small molecule targeted to inhibit activated NF-κB, a molecule that is activated from infancy in DMD and which is central to causing muscle damage and preventing muscle regeneration. Data on magnetic resonance imaging of the lower and upper leg muscles, physical function (including timed function tests) and muscle strength will be studied.

DETAILED DESCRIPTION:
Part A was a 1-week, open-label study to assess safety, tolerability, pharmacokinetics and biomarkers for three dose levels of edasalonexent and is now complete.

Part B was a randomized, double-blind, placebo-controlled, multiple dose study to evaluate the safety, efficacy, PK, and PD of edasalonexent over 12 weeks. Patients who participated in Part A also participated in Part B, along with newly enrolled patients. Patients received either edasalonexent 67 mg/kg/day, edasalonexent 100 mg/kg/day, or placebo in Part B. Part B is now complete.

Following completion of Part B, patients receive edasalonexent for 138 weeks in Part C, the open-label portion of the MoveDMD study. Patients on the 67 mg/kg/day treatment moved to the 100 mg/kg/day treatment. Patients on the 100 mg/kg/day treatment remained on the 100 mg/kg/day treatment. If clinically indicated, concomitant treatment with eteplirsen (Exondys 51™) may be acceptable in patients with amenable gene mutations during Part C after the patient has been exposed to edasalonexent for 6 months.

**Following completion of MoveDMD Part C, access to edasalonexent for trial participants will continue through the open-label extension study, GalaxyDMD.**

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from parent or legal guardian prior to participation and, for patients who are 7 years of age, written assent from patient
* Diagnosis of DMD based on a clinical phenotype with increased serum CK and the presence of a mutation in the dystrophin gene known to be associated with a DMD phenotype
* Ability to walk independently (assistive devices are permitted)
* Adequate immunization for influenza and varicella

Exclusion Criteria:

* Use of corticosteroids within prior 6 months of treatment initiation or planning to initiate steroid therapy within the next 6 months
* Other prior or ongoing significant medical conditions
* Exposure to another investigational drug (such as eteplirsen or idebenone) within 28 days prior to start of study treatment or ongoing participation in any other therapeutic clinical trial

  * Note: There are separate criteria for patients who participated in Part A versus newly enrolling patients. New patients must meet all of the Part A entry criteria to participate in Part B.

Patients who participated in Part A must meet the following criteria to participate in Part B:

* Completed Part A
* Continue to meet all of the Part A entry criteria, including an absence of safety concerns (however, patients may be ≥8 years of age)

There are no entry criteria for Part C; all patients who complete Part B will automatically continue in Part C

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01-12 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Los Angeles, California
  - Gainesville, Florida
  - Orlando, Florida
  - Portland, Oregon
  - Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 3-part, Phase 1/2, multi-centre study conducted at 5 study centers in United States.
Pre-assignment Details: A total of 32 patients were treated with edasalonexent in this study. 17 patients were enrolled in Part A and 16 completed 7 days of dosing, 1 patient screen failed due to inability to comply with study procedures and did not continue to Part B. A total of 31 patients (16 subjects from Part A and 15 New subjects who entered Part B) were enrolled in Part B, and all completed the 12 weeks of dosing. All 31 patients included in Part B enrolled in the open-label long-term extension phase, Part C.
Groups:
- Part A: Dose 1: Edasalonexent 33 mg/kg/day. Capsules taken by mouth two times per day
  Edasalonexent
- Part A: Dose 2; Part B: Dose 1; Part C: Dose 1: Edasalonexent 67 mg/kg/day. Capsules taken by mouth two times per day
  Edasalonexent
- Part A: Dose 3; Part B: Dose 2; Part C: Dose 2: Edasalonexent 100 mg/kg/day. Capsules taken by mouth three times per day
  Edasalonexent
- Part B: Placebo 1: Placebo 67 mg/kg/day Capsules taken by mouth two times per day
- Part B: Placebo 2: Placebo 100 mg/kg/day Capsules taken by mouth three times per day
Period: PartA(7 Day Open-Label Treatment Period)
Arm/Group | Part A: Dose 1 | Part A: Dose 2 | Part A: Dose 3 | Part B: Dose 1 | Part B: Dose 2 | Part B: Placebo 1 | Part B: Placebo 2 | Part C: Dose 1 | Part C: Dose 2
Started | 5 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Screen failure | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (12-week Double Blind)
Arm/Group | Part A: Dose 1 | Part A: Dose 2 | Part A: Dose 3 | Part B: Dose 1 | Part B: Dose 2 | Part B: Placebo 1 | Part B: Placebo 2 | Part C: Dose 1 | Part C: Dose 2
Started (It includes 16 Subjects who completed Part A and continued to Part B plus 15 New subjects who entered Part B) | 0 | 0 | 0 | 10 (4 New subjects plus 6 subjects who completed Part A) | 10 (4 New subjects plus 6 subjects who completed Part A) | 5 (3 New subjects plus 2 subjects who completed Part A) | 6 (4 New subjects plus 2 subjects who completed Part A) | 0 | 0
Completed | 0 | 0 | 0 | 10 | 10 | 5 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C (138-week, Open-label Treatment)
Arm/Group | Part A: Dose 1 | Part A: Dose 2 | Part A: Dose 3 | Part B: Dose 1 | Part B: Dose 2 | Part B: Placebo 1 | Part B: Placebo 2 | Part C: Dose 1 | Part C: Dose 2
Started (It has Subjects completed Part B) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 16
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Parent or Guardian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6

BASELINE CHARACTERISTICS:
Population: Safety population:
  Part A:The Safety Population was all patients who received at least 1 dose of IP in Part A
  Part B:The Safety Population was all patients who received at least 1 dose of IP in Part B.
  Active B or C Safety Population: The Safety Population was all patients who received at least 1 dose of active treatment in Part B and all patients who received placebo in Part B and at least 1 dose of active treatment in Part C.
Groups:
- Part A -CAT-1004 33 mg/kg/Day: Edasalonexent 33 mg/kg/day. Capsules taken by mouth two times per day
  Edasalonexent
- Part A - CAT-1004 67 mg/kg/Day; Part B - CAT-1004 67 mg/kg/Day: Edasalonexent 67 mg/kg/day. Capsules taken by mouth two times per day
  Edasalonexent
- Part A - CAT-1004 100 mg/kg/Day; Part B - CAT-1004 100 mg/kg/Day: Edasalonexent 100 mg/kg/day. Capsules taken by mouth three times per day
  Edasalonexent
- Part B: Overall Placebo: Placebo1:Placebo 67 mg/kg/day Capsules taken by mouth two times per day Placebo2: Placebo 100 mg/kg/day Capsules taken by mouth three times per day
- Total: Total of all reporting groups
Arm/Group | Part A -CAT-1004 33 mg/kg/Day | Part A - CAT-1004 67 mg/kg/Day | Part A - CAT-1004 100 mg/kg/Day | Part B - CAT-1004 67 mg/kg/Day | Part B - CAT-1004 100 mg/kg/Day | Part B: Overall Placebo | Total
Number analyzed (Participants) | 5 | 6 | 6 | 10 | 10 | 11 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analysis population are reported separately based on Part A and Part B.
  years
    Part A: number analyzed (Participants) | 5 | 6 | 6 | 0 | 0 | 0 | 17
    Part A | 5.2 (1.10) | 5.5 (0.55) | 5.7 (1.21) |  |  |  | 5.5 (0.94)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 10 | 10 | 11 | 31
    Part B |  |  |  | 5.97 (1.137) | 6.00 (1.165) | 6.34 (1.032) | 6.11 (1.086)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analysis population are reported separately based on Part A and Part B.
  Participants
    Part A: number analyzed (Participants) | 5 | 6 | 6 | 0 | 0 | 0 | 17
    Part A: Female | 0 | 0 | 0 |  |  |  | 0
    Part A: Male | 5 | 6 | 6 |  |  |  | 17
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 10 | 10 | 11 | 31
    Part B: Female |  |  |  | 0 | 0 | 0 | 0
    Part B: Male |  |  |  | 10 | 10 | 11 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analysis population are reported separately based on Part A and Part B.
  Participants
    Part A: number analyzed (Participants) | 5 | 6 | 6 | 0 | 0 | 0 | 17
    Part A: Hispanic or Latino | 0 | 0 | 1 |  |  |  | 1
    Part A: Not Hispanic or Latino | 4 | 6 | 5 |  |  |  | 15
    Part A: Unknown or Not Reported | 1 | 0 | 0 |  |  |  | 1
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 10 | 10 | 11 | 31
    Part B: Hispanic or Latino |  |  |  | 2 | 1 | 0 | 3
    Part B: Not Hispanic or Latino |  |  |  | 8 | 9 | 11 | 28
    Part B: Unknown or Not Reported |  |  |  | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analysis population are reported separately based on Part A and Part B.
  Participants
    Part A: number analyzed (Participants) | 5 | 6 | 6 | 0 | 0 | 0 | 17
    Part A: American Indian or Alaska Native | 0 | 0 | 0 |  |  |  | 0
    Part A: Asian | 0 | 0 | 0 |  |  |  | 0
    Part A: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  |  | 0
    Part A: Black or African American | 0 | 0 | 0 |  |  |  | 0
    Part A: White | 5 | 6 | 6 |  |  |  | 17
    Part A: More than one race | 0 | 0 | 0 |  |  |  | 0
    Part A: Unknown or Not Reported | 0 | 0 | 0 |  |  |  | 0
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 10 | 10 | 11 | 31
    Part B: American Indian or Alaska Native |  |  |  | 0 | 0 | 0 | 0
    Part B: Asian |  |  |  | 1 | 0 | 0 | 1
    Part B: Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0 | 1 | 1
    Part B: Black or African American |  |  |  | 0 | 1 | 0 | 1
    Part B: White |  |  |  | 9 | 9 | 9 | 27
    Part B: More than one race |  |  |  | 0 | 0 | 0 | 0
    Part B: Unknown or Not Reported |  |  |  | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: Analysis population are reported separately based on Part A and Part B
  Participants
    United States: Part A | 5 | 6 | 6 | 0 | 0 | 0 | 17
    United States: Part B | 0 | 0 | 0 | 10 | 10 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Lower Leg Composite of the MRI T2 Relaxation Time (LLC5-T2) - Part B
Description: The LLC5-T2 calculated from the unweighted average of the T2 relaxation times of all 5 lower leg muscles for each patient at each evaluation (the medial gastrocnemius, peroneals, soleus, tibialis anterior, and tibialis posterior muscles). Increases in LLC5-T2 relaxation time indicate muscle damage, inflammation, edema, and fat infiltration and are highly correlated with muscle fat
Time Frame: Baseline to Week 12
Population: Part B Full Analysis Population: The Full Analysis Population was a modified intent-to-treat population and consisted of all patients who received at least 1 dose of investigational product (IP) in Part B and had a valid baseline and at least 1 post baseline timed function test (TFT) or MRI efficacy assessment.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Part B - Placebo (Overall): Placebo 67 mg/kg/day Capsules taken by mouth two times per day
  Placebo 100 mg/kg/day Capsules taken by mouth three times per day
Arm/Group | Part B - CAT-1004 67 mg/kg/Day | Part B - CAT-1004 100 mg/kg/Day | Part B - Placebo (Overall)
Number analyzed (Participants) | 10 | 10 | 11
msec
  Baseline to Week 12 Endpoint - Soleus | 2.04 (3.179) | 1.26 (2.913) | 0.34 (2.380)
  Baseline to Week 12 Endpoint - Medial Gastrocnemius | 0.35 (2.410) | -0.16 (2.003) | 1.16 (2.517)
  Baseline to Week 12 Endpoint - Tibialis Anterior | -0.25 (2.558) | 0.01 (1.433) | 0.00 (1.878)
  Baseline to Week 12 Endpoint - Tibialis Posterior | 0.62 (1.107) | -1.05 (2.447) | -0.42 (2.716)
  Baseline to Week 12 Endpoint - Peroneal | 0.28 (2.764) | 0.63 (2.290) | 1.27 (1.630)

2. Secondary Outcome: Change From Baseline in the Speed of Completing the 10-meter Walk/Run Test (10MWT) at Week 12 - Part B and Part C
Description: The 10MWT determines the speed to walk a distance of 10 meters. The initial measurement was made in seconds and the speed of completing the test (i.e., calculated as the reciprocals of the time to complete; speed=1/time) is provided as the measure.
  For patients who are not able to complete the test, the speed of 0 will be imputed.
Time Frame: Baseline to Week 12
Population: The Active B or C Full Analysis Population consisted of the pooled patient populations of Parts B and C that received treatment in either part and had valid baseline and efficacy measurements.
Measure: Mean (Standard Deviation); unit: 10 meters/sec
Groups:
- Part C - CAT-1004 67 mg/kg/Day: Edasalonexent 67 mg/kg/day. Capsules taken by mouth two times per day
  Edasalonexent
- Part C - CAT-1004 100 mg/kg/Day: Edasalonexent 100 mg/kg/day. Capsules taken by mouth three times per day
  Edasalonexent
- Part B - Overall Placebo: Placebo 67 mg/kg/day Capsules taken by mouth two times per day
  Placebo 100 mg/kg/day Capsules taken by mouth three times per day
Arm/Group | Part C - CAT-1004 67 mg/kg/Day | Part C - CAT-1004 100 mg/kg/Day | Part B - Overall Placebo
Number analyzed (Participants) | 15 | 16 | 11
10 meters/sec | -0.0008 (0.01742) | -0.0041 (0.01584) | -0.0100 (0.01627)

3. Secondary Outcome: Change From Baseline in the Speed of Completing the 4-Stairs Climb Task at Week 12 - Part B and Part C
Description: The 4-stair climb test determines the speed to climb 4 standard steps. The initial measurement was made in seconds and the speed of completing the test (i.e., calculated as the reciprocals of the time to complete; speed=1/time) is provided as the measure.
  For patients who are not able to complete the test, the speed of 0 will be imputed.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 4 Stairs/Sec
Arm/Group | Part C - CAT-1004 67 mg/kg/Day | Part C - CAT-1004 100 mg/kg/Day | Part B - Overall Placebo
Number analyzed (Participants) | 15 | 16 | 11
4 Stairs/Sec | -0.0032 (0.07487) | -0.0046 (0.06223) | -0.0121 (0.06647)

4. Secondary Outcome: Change From Baseline in the Speed of Completing the Stand From Supine Task at Week 12 - Part B and Part C
Description: The stand from supine test determines the speed to stand from a supine position. The initial measurement was made in seconds and the speed of completing the test (i.e., calculated as the reciprocals of the time to complete; speed=1/time) is provided as the measure.
  For patients who are not able to complete the test, the speed of 0 will be imputed.
Time Frame: Baseline to Week 12
Population: Active B or C Full Analysis Population
Measure: Mean (Standard Deviation); unit: /Sec
Arm/Group | Part C - CAT-1004 67 mg/kg/Day | Part C - CAT-1004 100 mg/kg/Day | Part B - Overall Placebo
Number analyzed (Participants) | 15 | 16 | 11
/Sec | -0.0293 (0.04930) | -0.0042 (0.03890) | -0.0007 (0.05449)

5. Secondary Outcome: Safety and Tolerability Measured by Number of Treatment- Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs).
Description: A TEAE was any adverse event (AE) that started during or after the first dose of IP through the end of the safety follow-up period. Part B TEAEs were those that started on or after the first dose date in Part B through the date of Week 12 clinic dose. TEAEs for the Part C (Active B or C) analysis were those that started on or after the first dose date of active treatment in Part B or Part C. Drug related AEs included those marked as "Related" or "Possibly Related" to the study treatment.
Time Frame: Screening to Week 152
Population: Part A Safety Population (referred to in tables as All Dosed Patients) The Safety Population was all patients who received at least 1 dose of IP in Part A.
  Part B Safety Population: The Safety Population was all patients who received at least 1 dose of IP in Part B.
  Active B or C Safety Population: The Safety Population was all patients who received at least 1 dose of active treatment in Part B and all patients who received placebo in Part B and at least 1 dose of active treatment in Part C.
Measure: Count of Participants; unit: Participants
Groups:
- Part A - CAT-1004 33 mg/kg/Day: Edasalonexent 33 mg/kg/day. Capsules taken by mouth two times per day
  Edasalonexent
Arm/Group | Part A - CAT-1004 33 mg/kg/Day | Part A - CAT-1004 67 mg/kg/Day | Part A - CAT-1004 100 mg/kg/Day | Part B - CAT-1004 67 mg/kg/Day | Part B - CAT-1004 100 mg/kg/Day | Part B - Overall Placebo | Part C - CAT-1004 67 mg/kg/Day | Part C - CAT-1004 100 mg/kg/Day
Number analyzed (Participants) | 5 | 5 | 6 | 10 | 10 | 11 | 15 | 16
Participants
  Patients with any AEs after first dose | 2 | 5 | 5 | 0 | 0 | 0 | 0 | 0
  Patients with any AE related to study drug | 2 | 2 | 5 | 0 | 0 | 0 | 0 | 0
  Patients with any SAE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Patients with any AE leading to discontinuation from study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Patients with any TEAE | 0 | 0 | 0 | 9 | 8 | 10 | 15 | 16
  Patients with any drug-related TEAE | 0 | 0 | 0 | 5 | 7 | 1 | 8 | 11
  Patients with any TEAE leading to study drug discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Patients with drug-related TEAEs leading to study drug discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Upto 152 weeks
Description: Adverse events were collected from the time of signing the informed consent through study completion. A TEAE was an adverse event that started during or after the first dose of investigational product during Part B through the date of Week 12 clinic dose. At each level of summation (overall, system organ class, preferred term), patients reporting more than 1 AE were counted only once for the total incidence.
Arm/Group | Part A - CAT-1004 33 mg/kg/Day | Part A - CAT-1004 67 mg/kg/Day | Part A - CAT-1004 100 mg/kg/Day | Part B - CAT-1004 67 mg/kg/Day | Part B - CAT-1004 100 mg/kg/Day | Part B - Overall Placebo | Part C - CAT-1004 67 mg/kg/Day | Part C - CAT-1004 100 mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/10 | 0/10 | 0/11 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/10 | 1/10 | 0/11 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 2/5 | 5/6 | 5/6 | 9/10 | 8/10 | 9/11 | 15/15 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - CAT-1004 33 mg/kg/Day (N=5) | Part A - CAT-1004 67 mg/kg/Day (N=6) | Part A - CAT-1004 100 mg/kg/Day (N=6) | Part B - CAT-1004 67 mg/kg/Day (N=10) | Part B - CAT-1004 100 mg/kg/Day (N=10) | Part B - Overall Placebo (N=11) | Part C - CAT-1004 67 mg/kg/Day (N=15) | Part C - CAT-1004 100 mg/kg/Day (N=16)
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - CAT-1004 33 mg/kg/Day (N=5) | Part A - CAT-1004 67 mg/kg/Day (N=6) | Part A - CAT-1004 100 mg/kg/Day (N=6) | Part B - CAT-1004 67 mg/kg/Day (N=10) | Part B - CAT-1004 100 mg/kg/Day (N=10) | Part B - Overall Placebo (N=11) | Part C - CAT-1004 67 mg/kg/Day (N=15) | Part C - CAT-1004 100 mg/kg/Day (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Excessive eye blinking (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid rash (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 4 | 5 | 1 | 7 | 10
Faeces soft (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 2 | 0 | 3 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3 | 1 | 7 | 7
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 8
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 1 | 6 | 4
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 5
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 6
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 4 | 2 | 4 | 12 | 12
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0 | 5 | 3
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coagulation time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza B virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Emotional distress (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Impulsive behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Stubbornness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Negativism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep terror (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tic (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enuresis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 5 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pectus excavatum (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abasia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scarlet fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No